CLINICAL TRIAL: NCT06357130
Title: Gynaecological Care for Transgender People in France in 2024.
Acronym: GyneTrans
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/75
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Transgender Management Care
Keywords: Gynaecology; Gender-affirming hormonal therapy; Breast Cancer; Transgender; Contraception
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transgender: Transgender population in France, male to female and female to male.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A flyer with QR code leading to the online questionnaire will be sent to trans associations and healthcare networks for distribution to the target population.

SUMMARY:
To date, the transgender population, still poorly characterized, tends to increase. The impact of gender-affirming hormone therapy (GAHT) in this population remains poorly understood, and few data are published on the gynecological repercussions of such therapy. A recent literature review by a French team suggests gynecological follow-up procedures for transgender people.

DETAILED DESCRIPTION:
The hypothesis of this study is that transgender population in France does not have appropriate gynecological care, and the study would like to find out, directly from the people concerned, the current state of gynecological care for transgender people in France. To do this, ths study plan to send out a questionnaire to transgender people (via healthcare networks and also transgender associations) to ask them about their actual gynecological care and their knowledge of recommended gynecological care.

The aim is to set up a descriptive, declarative study based on a questionnaire created specifically for this work.

This project will use a questionnaire for transwomen people and another one for transmen people. Transgender people will be approached via Trans associations and healthcare networks. An online link to the questionnaire will be sent to trans associations and healthcare networks for distribution to the target population thanks to a flyer.

ELIGIBILITY:
Inclusion Criteria:

* French-speaking transgender person (transgender women or transgender men)
* age ≥18 years

Exclusion Criteria:

* age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Transgender people (male and female) will be approached via Trans associations (face-to-face and online) and the care networks in place at national level.
  An online link for completing the questionnaire will be sent to trans associations and healthcare networks for distribution to the target population via a paper or digital flyer.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of people aware of gynaecological recommendations. | 24 months after inclusion day
  Percentage of transgender people who know regular gynaecological recommendations in France, thanks to a homemade questionnaire

SECONDARY OUTCOMES:
Percentage of people aware of cancer risks | 24 months after inclusion day
  Overview of organized screening for gynaecological cancers and prostate cancer in the transgender population, thanks to a homemade questionnaire
Percentage of people aware of contraception in transgender male population | 24 months after inclusion day
  Overview of knowledge about contraception in the transgender male population,thanks to a homemade questionnaire.
Percentage of people aware of fertility and the impact of hormone treatments | 24 months after inclusion day
  Overview of knowledge about fertility and the impact of hormone treatments in the transgender population, thanks to a homemade questionnaire.
Percentage of people aware of gynaecological repercussions of masculinizing hormone treatment in transgender male population | 24 months after inclusion day
  Overview of our knowledge of the gynaecological repercussions of masculinizing hormone treatment in the transgender male population, thanks to a homemade questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Haut-Lévêque, Pessac, France